CLINICAL TRIAL: NCT04817085
Title: Prospective Multicenter, Randomized, Double-Masked, Controlled Trial to Evaluate Clinical Utility and Safety of the Visant Medical Canalicular Device in Subjects Who Are Candidates for Occlusion With Punctal or Canalicular Plugs
Brief Title: An Evaluation of the Clinical Utility and Safety of the Visant Medical Canalicular Plug
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visant Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-348-CSP
Record Dates: First submitted 2020-12-02; First posted 2021-03-25 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All study subjects will receive treatment. Study subjects will be randomized (2:1 ratio) with 2 subjects randomized to receive the Visant Medical Canalicular Plug for every 1 subject randomized to receive the commercially available canalicular plug.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be masked to their assignment to either the treatment or control group. Clinical personnel who perform clinical assessments will also be masked to the subjects' assignment to either the treatment or control group ("masked evaluators"). The eye care professional who inserts the test and control devices will not be masked and will not be eligible to perform follow-up evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Visant Medical Canalicular Plug (Experimental): Bilateral placement of the Visant Canalicular Plug inserted on Day 1
  Interventions: Device: Visant Medical Canalicular Plug
- Commercially available canalicular plug (Active Comparator): Bilateral placement of commercially available canalicular plug inserted on Day 1
  Interventions: Device: Commercially available canalicular plug

INTERVENTIONS:
Device: Visant Medical Canalicular Plug — Plug is inserted into the inferior canaliculi and assessed for 6 months
  Arms: Visant Medical Canalicular Plug
Device: Commercially available canalicular plug — Plug is inserted into the inferior canaliculi and assessed for 6 months
  Arms: Commercially available canalicular plug

SUMMARY:
This study is designed to evaluate the clinical utility and safety of the Visant Medical Canalicular Plug compared to a commercially available canalicular plug.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the clinical utility and safety of the Visant Medical Canalicular Plug compared to a commercially available canalicular plug over 6 months of subject follow-up.

Study subjects who are eligible for enrollment and have provided written informed consent will be randomized in a 2:1 ratio (i.e., 2 subjects randomized to the Visant Medical Canalicular Plug for every 1 subject randomized to a commercially available canalicular plug). All study subjects will be treated bilaterally with plugs placed in the inferior canaliculi.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty-two (22) years of age or older
2. BCDVA of 20/40 or better in each eye
3. Both eyes with a baseline Schirmer's test with anesthetic ≤ 10 mm/5 minutes
4. Presence of corneal staining in both eyes in any of the 5 areas defined by the NEI/Industry Workshop Scale
5. Baseline OSDI score of at least 23 with no more than 3 responses of "not applicable"
6. Patent bilateral lacrimal drainage system as demonstrated by punctal irrigation
7. If female, subject must be post-menopausal, medically sterile (e.g hysterectomy, bilateral tubal ligation, bilateral oophorectomy) or have negative urine pregnancy test (UPT) on Day 0 of the study and agree to utilize a medically acceptable form of contraception over the course of the study
8. Willing and able to sign informed consent and HIPAA authorization, follow study instructions, and complete all study visits.

Exclusion Criteria:

1. Use of ophthalmic cyclosporine (Restasis) within 6 months or lifitegrast (Xiidra) within 3 months prior to Day 0 in either eye
2. History of surgical punctal occlusion (e.g., cautery), canalicular infection or canalicular surgery in either eye
3. Corneal transplant in either eye
4. Ocular surgery (such as cataract surgery or LASIK) in either eye within six months of the Baseline Visit
5. A systemic condition or disease not stabilized or judged by the investigator to be incompatible with participation in the study (e.g. current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease)
6. The history or presence of any ocular disorder or condition in either eye that, in the opinion of the investigator, would interfere with the interpretation of the study results (e.g., significant corneal or conjunctival scarring, pterygium or nodular pinguecula; current ocular infection (except mild blepharitis), conjunctivitis or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; history of ocular herpetic infection; evidence of keratoconus; lid or lacrimal cancer
7. Active severe systemic allergy, seasonal allergies, rhinitis or sinusitis requiring treatment (i.e., antihistamines, decongestants, oral or aerosol steroids)
8. Use of steroids, including administration by systemic or topical ocular routes (dermatologic steroids not applied to the eyelids and inhaled steroids are allowed)
9. Participation in a clinical trial during the past 30 days
10. Women who are pregnant, planning a pregnancy, or nursing at study entry

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Mean change in Schirmer's score from baseline to Month 3 compared to commercially available plug | 3 months
  Non-inferiority hypothesis. Higher Score using this continuous variable equates to larger tear film

SECONDARY OUTCOMES:
Proportion of responders achieving improvement from Baseline in Ocular Surface Disease Index (OSDI) score by a Minimal Clinically Important Difference (MCID). | 3 months
  Non-inferiority hypothesis. Scale of 0-100. Lower OSDI score means fewer symptoms.
Mean change in tear meniscus height from baseline | Month 3
  Null hypothesis of no improvement from baseline. Larger measurement equates to larger tear film.
Mean change in OSDI score from baseline | Month 3
  Null hypothesis of no improvement from baseline. Non-inferiority hypothesis. Scale of 0-100. Lower OSDI score means fewer symptoms.
Mean change in corneal staining score from baseline (NEI workshop scale) | Month 3
  Null hypothesis of no improvement from baseline. Scale is 0-15. More staining is associated with more severe dry eye.
Mean change in tear meniscus height from baseline | Month 6
  Null hypothesis of no improvement from baseline. Larger measurement equates to larger tear film.
Mean change in OSDI score from baseline | Month 6
  Null hypothesis of no improvement from baseline. Non-inferiority hypothesis. Scale of 0-100. Lower OSDI score means fewer symptoms.
Mean change in corneal staining score from baseline (NEI workshop scale) | Month 6
  Null hypothesis of no improvement from baseline. Scale is 0-15. More staining is associated with more severe dry eye.
Mean change in tear break up time from baseline | Month 3
  Null hypothesis of no improvement from baseline. Increased time equates to more stable tear film
Mean change in Schirmer score from baseline | Month 6
  Null hypothesis of no improvement from baseline. Higher Score using this continuous variable equates to larger tear film
Mean change in tear break up time from baseline | Month 6
  Null hypothesis of no improvement from baseline. Increased time equates to more stable tear film

CONTACTS AND LOCATIONS:
Overall Officials: Roger Albright, Study Director — Ora Clinical Research Organization
Locations (5):
- United States (5):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Eye Research Foundation, Inc., Newport Beach, California
  - Andover Eye Associates, Andover, Massachusetts
  - Piedmont Eye, Inc., Lynchburg, Virginia
  - See Clearly Vision, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No